CLINICAL TRIAL: NCT03169621
Title: Diagnosis of Chronic Endometritis in Endometrial Fluid Using Molecular Techniques to Improve the Outcomes of Assisted Reproductive Treatments
Acronym: ChEndometritis
Status: Terminated | Type: Observational
Why Stopped: Low patient enrolment during the recruiting period
Sponsor: Igenomix (Industry)
Collaborators: Instituto de Investigacion Sanitaria INCLIVA (Other); University of Valencia (Other)
Responsible Party: Sponsor
Other Study IDs: IGX1-ECR-CS-17-01
Record Dates: First submitted 2017-05-19; First posted 2017-05-30 (Actual); Last update posted 2019-03-26 (Actual); Status verified 2018-08

CONDITIONS: Chronic Endometritis
Keywords: Chronic Endometritis; Endometrial pathogens; Microbiological diagnosis; Next Generation Sequencing; Metagenomics; Endometrial receptivity

STUDY DESIGN:
Observational Model: Other | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — DNA will be analyzed in the endometrial fluid. These samples will be completely exhausted during the analysis.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Patients with RIF: Patients with repeated implantation failure (RIF) with indication of hysteroscopy within normal clinical practice, who will undergo FIV or ICSI and embryo transfer within their assisted reproduction treatment (ART).
  Interventions: Procedure: Endometrial Biopsy and endometrial fluid collection

INTERVENTIONS:
Procedure: Endometrial Biopsy and endometrial fluid collection — On day 5 of the Hormonal Replacement Therapy (after 5 days of progesterone administration), the doctor will perform endometrial fluid aspiration (EF) followed by an endometrial biopsy (EB) the same day of hysteroscopy that is performed as usual clinical practice. EF sample will be analyzed by molecular techniques (Next Generation Sequencing) for the detection of infectious agents and the EB sample will be divided into three parts, one of them will be used for molecular analysis (as control of the bacterial content present in the EF) and the others will be used for microbiological analysis and histological techniques respectively.
  The Assisted Reproductive Treatment (ART) will be performed once the specialist considers it appropriated according to the clinical standard practice and the reproductive rates will be correlated with the diagnosis of CE comparing the results of ART before and after its diagnosis of CE.

SUMMARY:
Chronic endometritis (CE) is a persistent inflammation of the endometrial lining caused by the infection of the uterine cavity mainly by bacterial pathogens. It is known that CE can produce implantation failure, recurrent abortion and preterm labor. The study hypothesis is that patients who have repeated implantation failures (RIF) despite transferring good quality and normal embryos, diagnosed by preimplantation Genetic Diagnosis (PGD), into a receptive endometrium, diagnosed by Endometrial Receptivity Analysis (ERA), may present asymptomatic CE, being the altered endometrium the main cause of these implantation failures.

The current diagnosis of CE is the microbiological culture of endometrial biopsy samples. Alternatively, examination of the uterine cavity by hysteroscopy is effective at 93.4%. However, both methods have limitations, such as the time needed to obtain the diagnosis, the economic cost of the tests, the possibility of detecting microorganisms in culture etc. For these reasons, the developing of a simple, fast, cheap and minimally invasive diagnostic tool for CE patients subjected to IVF treatments is expected. It would be very useful in order to establish a specific treatment and improve pregnancy rates in infertile patients. For this reason, the bacterial DNA present in the endometrial fluid samples will be obtained and the identification of the causative pathogens of CE will be done by sequencing (NGS) and/or quantitative PCR with specific oligonucleotides for the most common bacteria causing CE. The validation of this new method will be performed by comparison with the microbiological diagnosis of those same patients.

DETAILED DESCRIPTION:
On day 5 of the Hormonal Replacement Therapy (after 5 days of progesterone administration), coinciding with the day of hysteroscopy indicated by the physician according to the routine clinical practice, samples of endometrial fluid (EF) and endometrial biopsy (EB) of patients with RIF will be obtained. These samples will be used for the diagnosis of CE by both classic and molecular methods. Specifically, EF sample will be analyzed by molecular techniques using Next Generation Sequencing (NGS) for the detection of infectious agents. EB sample will be divided into three parts, one of them will be used for molecular analysis (as control of the bacterial content present in the EF), another part will be subjected to microbiological analysis and the third part will be analyzed using histological techniques. In this way, comparisons will be made between the different diagnostic methods of CE in the two sample types (EF and EB) and the efficacy values of the new diagnostic test (sensitivity, specificity, positive and negative predictive values and Receiving Operating Characteristic curves) will be obtained using the microbiological diagnosis as a reference (gold standard method).

Patients with a negative outcome for CE (approximately 40%) will continue with the expected assisted reproduction treatment (ART) according to the clinic's standard protocol and patients with a positive outcome for CE (approx. 60%) will receive antibiotic treatment according to usual clinical practice (time and type of antibiotic will be different according to the microbiological diagnosis). Once this treatment is completed, the improvement of these patients will be confirmed obtaining a second sample of EF and EB. The Assisted Reproductive Treatment (ART) will be performed once the specialist considers it appropriated.

Finally, reproductive rates will be correlated with the diagnosis of CE. Therefore, an observational analytical study, in which a comparison of the ART results before and after its diagnosis of CE, will be carried out. The reproductive impact of an altered endometrial microbiota will be assessed analyzing the implantation rates, pregnancy and ongoing pregnancy.

ELIGIBILITY:
Inclusion Criteria:

* Patients who provide their written informed consent after having been informed of the all study aspects.
* IVF or ICSI cycles with own oocytes, with blastocyst transfer (day 5 or 6 of stage development).
* Women with age comprised between 18 and 38 years (both included).
* Body mass index: 18.5 - 30 km/m2 (both included)
* Adequate ovarian reserve > 8 antral follicles (RFA) and/or Antimüllerian hormone (HAM)> 1 ng / mL.
* Concentration of spermatozoa > 2 million sperm/ml.

Exclusion Criteria:

* Congenital or acquired uterine pathologies.
* Endometriosis.
* Patients with IUDs in the last 3 months.
* Patients who have taken prescribed antibiotic treatment in the last 3 months.
* Any disease or medical condition that could be unstable or could endanger the security of the patient and her compliance in the study.

Ages: 18 Years to 38 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Study Population: Patients with repeated implantation failure with indication of hysteroscopy within normal clinical practice, who will undergo FIV or ICSI and embryo transfer within their assisted reproduction treatment at our center (Hospital Clínico Universitario de Valencia) .
Sampling Method: Non-Probability Sample
Enrollment: 5 (Actual)
Dates: Start 2017-04-27 (Actual); Primary Completion 2018-06-26 (Actual); Study Completion 2019-02-13 (Actual)

PRIMARY OUTCOMES:
Developing of a new non invasive diagnosis test by Next Generation Sequencing (NGS) analysis for patients diagnosed with chronic endometritis (CE). | 24 months
  DNA analysis by NGS using endometrial fluid for the CE diagnose.

SECONDARY OUTCOMES:
To compare the diagnose of CE, determined by classical and molecular methods measured by NGS, in both types of samples analyzed (endometrial fluid and endometrial biopsy). | 24 months
  Endometrial fluid will be used for the DNA analysis by NGS and endometrial biopsy will be used for the classical diagnosis ((microbial culture, histology and hysteroscopy).
Qualitative study of the endometrial microbiome by classical and molecular methods in order to determine their influence in the CE diagnose. | 24 months
  To determine the identity of pathogenic bacteria measured by NGS that could establish endometrial infection.
Quantitative study of the endometrial microbiome by classical and molecular methods in order to determine their influence in the CE diagnose. | 24 months
  To determine the minimal amount of pathogenic bacteria measured by NGS that could establish endometrial infection.
Relationship between the implantation rate and the diagnosis of CE, by molecular and classical methods, in patients undergoing assisted reproduction treatments (ART). | 6 weeks
  Implantation rate is defined as the number of gestational sacs observed by vaginal ultrasound per number of transferred embryos in the 6th gestational week.
Relationship between the ongoing pregnancy rate per embryo transfer and the diagnosis of CE, by molecular and classical methods, in patients undergoing assisted reproduction treatments (ART). | 5 months
  Ongoing pregnancy rate is defined as the number of ongoing pregnancies after the 20th gestational week per total number of embryo transfers performed.
Relationship between the live birth rate and the diagnosis of CE, by molecular and classical methods, in patients undergoing assisted reproduction treatments (ART). | 9 months
  Live birth rate is defined as the number of the total live births per total number of embryo transfers performed.

CONTACTS AND LOCATIONS:
Overall Officials: Carlos Simón, MD PhD, Study Chair — Igenomix; Gemma Arribas, MD PhD, Principal Investigator — Hospital Clínic Universitari
Locations (1):
- Hospital Clínic Universitari de Valencia - INCLIVA, Valencia, Spain

IPD SHARING:
Plan to Share IPD: No